CLINICAL TRIAL: NCT04786249
Title: Impact of Rapid Screening for COVID-19 in Delocalized Biology in the Emergency Department
Acronym: DELOCOVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DELOCOVID
Record Dates: First submitted 2021-03-05; First posted 2021-03-08 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: Rapid test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19), caused by SARS-CoV-2, first appeared in China, and then spread around the world. In December 2019, a group of patients with pneumonia of unknown origin were infected after exposure to the market in Wuhan, Hubei province, China. Very quickly, a new coronavirus was isolated from a sample of a patient's lower respiratory tract and the entire virus genome was sequenced. This new coronavirus, named Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) for its genetic homology with SARS-CoV-2, has shown worldwide expansion. Thus, on January 30, 2020, the World Health Organization (WHO) announced the COVID-19 epidemic as a threat to public health at the international level, then, in March 2020, the global situation degenerated into a pandemic. . Johns Hopkins University has reported more than 7,600,000 cases of infections and more than 427,000 deaths as of June 13, 2020. Due to the rapid progression of the COVID-19 pandemic and the limited capacity of molecular laboratory tests, the concept of delocalized molecular tests appears to be relevant. Indeed, the urgent need to increase testing for COVID-19 has been clearly identified as an essential part of the strategy to combat the coronavirus worldwide. In fact, COVID-19 represents a major public health problem currently causing a rapidly increasing number of infections and significant morbidity and mortality worldwide. As of July 1, 2020, more than 10 million people worldwide have been infected with SARS-CoV-2. As of December 20, 2020, this tally is 76,624,363 cases of contamination and 1,690,658 deaths following Johns Hopkins University

DETAILED DESCRIPTION:
Early detection with a sensitive technique of COVID-19 is essential to ensure rapid and appropriate patient management, to contain the epidemic and to better understand the global epidemiology of the virus. This detection will intensify in the coming months due to the start of the school year and university as well as the economic recovery. Until now, laboratory diagnostics have relied primarily on the amplification and detection of viral gene sequences in upper respiratory tract samples performed in a centralized laboratory. A new test (Abbott ID NowTM COVID-19) is available on the market. This test is the first in France to be able to be carried out in a delocalized medical biology examination (DMBE) and makes it possible to return a result in less than 15 min directly in the clinical department. The speed of this technique is based on the use of isothermal gene amplification. The investigators will be the first to evaluate it in France in delocalized biology.

The improvement in diagnostic technique, concomitant with the development of knowledge on the pathophysiology and specific therapies, has been accompanied by better therapeutic management of patients with Covid19. To date, dexamethasone represents the first class of drugs proven to be effective in reducing mortality from COVID-19 in patients with severe disease. Anticoagulant treatment at a prophylactic dose in hospitalized patients or at risk for the severe form, and at a curative dose for severe forms is also the subject of strong recommendations due to the high incidence of venous and arterial thromboembolic events in these patients. It is also recommended that the use of broad-spectrum antibiotics be reserved for patients with radiological abnormalities compatible with bacterial superinfection and / or requiring oxygen therapy greater than or equal to 6 liters / min.

In France, systematic screening for SARS-CoV-2 infection in the emergency room before hospitalization, an operating room, or transfer to another establishment. At GhPSJ, the reference RT-PCR technique Simplexa ™ COVID-19 Direct assay has been used routinely since July 2020 by the microbiology laboratory. It allows a result rendering in a minimum delay of 50 minutes. Since September 7, 2020, the prescription of an RT-PCR is systematically associated with a dedicated computerized questionnaire on the DxCare® software completed by the emergency physician. It collects the reason for prescribing RT-PCR: "diagnostic suspicion", "bed management", "preoperative screening", or "screening for transfer to another establishment"; the patient's lifestyle; the symptomatic or asymptomatic nature and the duration of the symptoms. Since October 22, 2020, the DMBE with the Test ID NowTM COVID-19 has been installed and implemented in the Emergency Department. It is used by the trained and authorized Emergency Nursing team for any patient having a prescription for RT-PCR Sars-CoV-2 by the emergency physician.

The investigators wish to verify the hypothesis that obtaining the rapid diagnosis of Sars-CoV-2 infection by DMBE in the emergency room (Test ID NowTM COVID-19) makes it possible to optimize the organizational and medical management of emergency room patients having a Sars-CoV-2 RT-PCR test. In the literature, there is no study available evaluating the impact of a rapid examination in delocalized biology on the medical management of patients in an emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient presenting to the emergency unit of the GhPSJ and for whom a PCR examination is prescribed by the emergency doctor in charge of the patient
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of their data for this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency unit of the GhPSJ and for whom a PCR examination is prescribed by the emergency doctor in charge of the patient during the two periods of 7 weeks:
  * Period 1 (weeks 37 to 43 of the year 2020): RT PCR SARS-CoV-2 was carried out in the microbiology laboratory
  * Period 2 (44 to 50 of the year 2020): diagnosis of SARS-CoV-2 infection with the ID Now ™ technique in emergencies in DMBE with respect for the standards and recommendations of delocalized biology.
  The number of patients included will be 1200 per period.
Sampling Method: Non-Probability Sample
Enrollment: 2488 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of a short delay in delivering results in delocalized biology on the emergency medical care time, in comparison with the reference method by RT-PCR at the central laboratory of microbiology | Day 1
  Time of medical care in the emergency department corresponding to the time between the first medical contact (time stamp of the medical observation traced in DxCare®) and the patient's discharge from the Emergency Department (time stamp of the stay in DxCare®)

SECONDARY OUTCOMES:
Evaluate the impact of the rapid result in DMBE in comparison with the reference method on the final orientation of the patient | Day 1
  Number of returns home and the number of hospitalizations in conventional services and intensive care.
Evaluate the impact of the rapid result in DMBE in comparison with the reference method on the bed management | Day 1
  Number of admissions in single and double rooms
Evaluate the impact of the rapid result in DMBE in comparison with the reference method on the number of additional examinations carried out and their deadline | Day 1
  Number of blood tests, ECG, chest X-ray, chest CT scan without injection, pulmonary CT angiography
Evaluate the impact of the rapid result in DMBE in comparison with the reference method on the prescriptions and the timeframe for the implementation of specific therapies against Covid-19 in hospitalized patients | Day 1
  Introduction of corticosteroid therapy and anticoagulation
Evaluate the impact of the rapid result in DMBE in comparison with the reference method on the prescription of antibiotic treatments | Day 1
  Number of antibiotic treatments
Compare the primary endpoint for two subgroups of patients according to their treatment schedule | Day 1
  Number of patients who had a PCR prescription by the day medical team between 8:31 a.m. and 6:30 p.m. and those who had a PCR prescription by the on-call medical team between 6:31 p.m. and 8:30 a.m.
Evaluate the level of satisfaction and the feelings of the medical and paramedical teams of the Emergency Department regarding the DMBE Test ID Now ™ COVID-19 and its impact | Day 1
  Staff questionnaire (satisfied or not satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude NGUYEN, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Gerlier C, Pilmis B, Ganansia O, Le Monnier A, Nguyen Van JC. Clinical and operational impact of rapid point-of-care SARS-CoV-2 detection in an emergency department. Am J Emerg Med. 2021 Dec;50:713-718. doi: 10.1016/j.ajem.2021.09.062. Epub 2021 Sep 28. PMID 34879491